CLINICAL TRIAL: NCT05856240
Title: Targeted Group-based Psychotherapy to Address Emotional Stress in at Risk ICU Survivors: A Pilot Feasibility Study
Brief Title: Targeted Group-based Psychotherapy to Address Emotional Stress in at Risk ICU Survivors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Personnel no longer available to begin study
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Katherine Berg, Assistant Professor, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023P000087
Record Dates: First submitted 2023-04-24; First posted 2023-05-12 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Post Intensive Care Syndrome; Anxiety; Traumatic Stress; Depression
MeSH Terms: conditions — postintensive care syndrome; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group-Based Psychological Intervention (Experimental): Single-arm feasibility trial, so all participants will receive the intervention.
  Interventions: Behavioral: Managing Stress & Emotions Group (MSEG)

INTERVENTIONS:
Behavioral: Managing Stress & Emotions Group (MSEG) — The intervention consists of 6, 90-minute weekly sessions and includes the following components: providing education about psychological and emotional reactions to stress, introducing and practicing coping skills (e.g., mindfulness, emotional awareness, flexible thinking, behavioral modification), decreasing psychological avoidance using emotional exposure, and facilitating group support and discussion (see De Paul & Caver, 2021 for original protocol description).

SUMMARY:
This study is a pilot clinical trial to assess the feasibility of implementing a group-psychotherapy intervention to modify emotional stress (e.g., anxiety, depression, post-traumatic stress) following ICU hospitalization

DETAILED DESCRIPTION:
Psychological symptoms and emotional distress, including anxiety, depression, and posttraumatic stress, are common problems among patients discharged from the intensive care unit (ICU). The presence of psychological distress is associated with poor medical adherence, slower recovery, and reduced quality of life in this patient population. There is a lack of research on evidence-based interventions to address mental health symptoms in ICU patients post-hospitalization. Researchers have recently highlighted the potential utility of peer support/group interventions in the post-ICU recovery process; however, they have yet to be widely tested in interventional trials, and their feasibility and acceptability in the post-ICU population have yet to be demonstrated in a research study. Thus, the purpose of this study is to adapt and deliver a 6-session group-based psychological intervention for post-ICU patients in a single-arm, non-randomized interventional study. Patients' symptoms will be assessed at baseline, post-intervention, and 3-month follow-up. The primary aim of the study is to assess the feasibility and acceptability of the group intervention in the post-ICU patient population. Secondarily, changes in patients' emotional distress will be examined to assess for the impact of the intervention on patients' symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18 years
* ICU stay of at least 3 days
* Access to a smartphone, laptop, or computer and able to participate in a meeting via a virtual platform
* Montreal Cognitive Assessment (MoCA)-BLIND score of at least 18
* English fluency
* Screening questionnaires consistent with clinically significant depression OR anxiety (Hospital Anxiety and Depression Scale-Depression [HADS-D] OR HADS-Anxiety [HADS- A] score of >7) OR Post-traumatic Stress (PTSD Checklist-Civilian Version [PCL-C] score of ≥ 30)
* Resides in the state of Massachusetts.

Exclusion Criteria:

* Unable or unwilling to participate in 6 weekly sessions of group therapy
* Permanent or severe cognitive impairment severe enough to impede participation (as assessed via the MMSE).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment | Baseline
  This will be determined by reporting the number of patients who meet study criteria who agreed to participate.
Adherence to sessions (acceptability) | At 6 weeks (immediately at end of intervention sessions)
  This will be determined by reporting the number of intervention sessions completed by each participant.
Feasibility of data collection at post-treatment | At 6 weeks (immediately at end of intervention sessions)
  This will be determined by reporting the number of participants who provide post-treatment data.
Feasibility of data collection at follow-up | At 3 months follow-up
  This will be determined by reporting the number of participants who provide follow-up data.
Client Satisfaction Questionnaire | At 6 weeks (immediately at end of intervention sessions)
  This measure assesses participants' satisfaction with the intervention (participant ratings of 1 to 4, higher scores indicate higher satisfaction).
Credibility and Expectancy Questionnaire | Baseline
  This measure assesses participants' expectations and beliefs that the intervention will be helpful (Participant ratings of 1 to 9, higher scores indicate higher beliefs that the intervention will be helpful).

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System-29 (PROMIS-29)- Anxiety | Change from Baseline to immediately Post-Intervention (at 6 weeks), and from Baseline to to 3-months Follow-up
  This sub-scale of the PROMIS measure assesses participants' anxiety symptoms (Participant ratings of 1 to 5, higher ratings indicate greater anxiety symptoms).
Patient-Reported Outcomes Measurement Information System-29 (PROMIS-29)- Depression | Change from Baseline to immediately Post-Intervention (at 6 weeks), and from Baseline to to 3-months Follow-up
  This sub-scale of the PROMIS measure assesses participants' depression symptoms (Participant ratings of 1 to 5, higher ratings indicate greater depression symptoms).
PTSD Checklist-Civilian Version (PCL-C) | Change from Baseline to immediately Post-Intervention (at 6 weeks), and from Baseline to to 3-months Follow-up
  This measure assesses participants' PTSD symptoms (Participant ratings of 1 to 5, higher ratings indicate greater PTSD symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Katherine M Berg, MD, Principal Investigator — Beth Israel Deaconess Medical Center

IPD SHARING:
Plan to Share IPD: No